CLINICAL TRIAL: NCT01247961
Title: Intravenous Dexamethasone for the Early Treatment of Mild Acute Pancreatitis: A Double-Blind, Randomized, Placebo Controlled Trial
Brief Title: Early Treatment With Dexamethasone in Mild Acute Pancreatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bechien Wu, MD, MPH, Physician, Center for Pancreatic Disease, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P-002192
Record Dates: First submitted 2010-11-19; First posted 2010-11-25 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Patients With Acute Pancreatitis
MeSH Terms: interventions — dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 mg intravenous dexamethasone (Experimental): Subjects randomized to intervention arm will receive single dose of 10 mg intravenous dexamethasone.
  Interventions: Drug: Dexamethasone acetate
- Placebo (Placebo Comparator): Equal volume of normal saline administered as a single intravenous dose at enrollment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone acetate — 10 mg intravenous given as single administration with optional repeat dose after 36 hours.
  Arms: 10 mg intravenous dexamethasone
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
This pilot trial will evaluate the following in patients with acute pancreatitis:

1. Safety profile of early treatment with intravenous dexamethasone
2. Impact of dexamethasone on systemic inflammation in patients with acute pancreatitis
3. Provide preliminary data on potential impact of early treatment with steroids on clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years
* Diagnosis of acute pancreatitis confirmed by at least 2 of the following:

  1. Typical epigastric abdominal pain
  2. Elevation amylase/lipase >3 times upper limit normal and/or
  3. Confirmatory findings on cross-sectional imaging
* Enrollment within 8 hours of presentation

Exclusion Criteria:

* Class II or greater NYHA heart failure
* Oxygen dependent COPD
* Chronic kidney disease>stage 2
* Cirrhosis
* Existing necrosis on abdominal CT
* Organ dysfunction prior to enrollment
* Sepsis
* Acute respiratory distress syndrome
* Malignancy not in remission for at least 5 years
* Active drug use
* Known allergy to dexamethasone
* Altered mental status
* Insulin-requiring diabetes
* Abdominal surgery within 60 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammation (measured by c-reactive protein level) | 48 hours
  C-reactive protein (CRP) is a well-established inflammatory prognostic marker in acute pancreatitis. Primary comparison will be between median CRP levels at 48 hours between treatment arms.

SECONDARY OUTCOMES:
Safety parameters | 72 hours post-randomization
  We will monitor for incidence of malignant hyperglycemia (blood sugar>400 mg/dL), psychosis or culture-documented infectious complications.
Composite clinical outcome | Up to 14 days from hospital admission
  A composite clinical endpoint including development of either 1) pancreatic necrosis, 2) persistent organ dysfunction defined according to Atlanta symposium criteria 3) requirement for treatment in an intensive care unit and/or 4) development of culture-documented infection will be used to evaluate impact of treatment with dexamethasone on clinical outcomes in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Bechien U Wu, MD, MPH, Principal Investigator — Center for Pancreatic Disease, Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States